CLINICAL TRIAL: NCT07121439
Title: The Efficacy and Safety of a Combined Serum Containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and Hydroxyethylpiperazine Ethane Sulfonic Acid Following Low-Fluence Q-Switched Nd:YAG 1064 nm Laser Treatment for Melasma and Post-Acne Hyperpigmentation Therapy
Brief Title: Efficacy and Safety of a Combined Serum Containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, Sp.D.V.E., Subsp.D.K.E. - Head of Cosmetic Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: melab3
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Melasma; Post-acne Hyperpigmentation
MeSH Terms: conditions — Melanosis | interventions — Niacinamide; Hyaluronic Acid; HEPES

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): Participants receive the test serum containing Melasyl™, Niacinamide 10%, Hyaluronic Acid, and HEPES every morning and night, plus SPF >30 sunscreen every morning.
  Interventions: Drug: a combination serum containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES
- control (Active Comparator): Participants receive 2% hydroquinone cream at night and SPF >30 sunscreen every morning.
  Interventions: Drug: 2% hydroquinone cream

INTERVENTIONS:
Drug: a combination serum containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES — Subjects were randomized to receive a combination serum The combination serum contained Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES. applied twice daily, following QS-Nd:YAG 1064 nm low-fluence laser treatment. Clinical evaluations were conducted at baseline and at Weeks 1, 2, and 4 post-laser to assess pigmentation improvement, erythema, and overall skin condition.
  Arms: treatment
Drug: 2% hydroquinone cream — Subjects were randomized to received 2% hydroquinone cream, applied once daily at night, following QS-Nd:YAG 1064 nm low-fluence laser treatment. Clinical evaluations were conducted at baseline and at Weeks 1, 2, and 4 post-laser to assess pigmentation improvement, erythema, and overall skin condition.
  Arms: control

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of a combination serum containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES when used as a moisturizer after QS-Nd:YAG 1064 nm low-fluence laser treatment for melasma and post-acne hyperpigmentation.

The study aims to answer the following main questions:

* Does the combination serum reduce hyperpigmented lesions after laser treatment for melasma and post-acne hyperpigmentation?
* Does the serum improve skin hydration following laser therapy for melasma?
* Is the combination serum safe for use after laser treatment, without causing irritation or adverse effects?

Participants will be female patients aged 18-60 years, clinically diagnosed with melasma or post-acne hyperpigmentation (skin types IV and V), who visit the Dermatology & Venereology Outpatient Clinic for QS-Nd:YAG 1064 low-fluence laser treatment. All participants will have undergone a 2-week priming period using either 2% hydroquinone cream or the test serum prior to laser treatment. Written informed consent is required.

Participants will be randomly assigned to receive either the test serum or 2% hydroquinone cream based on a coded allocation. The product will be applied twice daily after facial cleansing, and sunscreen will be used 15 minutes before outdoor activities. Treatment lasts for 2 weeks, with participants recording application times and any adverse effects in a diary. Evaluations-including facial photography, mMASI, mexameter, dermoscopy, Wood's lamp, and PAHPI-will be conducted at baseline and at 1, 2, and 4 weeks post-laser. Erythema and subjective assessment (VAS) will be performed 15 minutes after the laser procedure.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial aimed at evaluating the efficacy and safety of a combination serum containing Melasyl™, 10% Niacinamide, Hyaluronic Acid, and HEPES as a moisturizer following QS-Nd:YAG 1064 nm low-fluence laser treatment in patients with melasma and post-acne hyperpigmentation. Medical history, physical examination, and laser procedures will be performed at the Dermatology and Venereology Clinic of Gatot Soebroto Central Army Hospital (RSPAD), Jakarta. Participants will be stratified based on their condition (melasma or post-acne hyperpigmentation) and randomly allocated using coded assignment into two groups. Group 1 (control) will receive 2% hydroquinone cream applied nightly, along with sunscreen with SPF >30 applied every morning. Group 2 (intervention) will receive the combination serum applied twice daily (morning and evening), along with the same SPF >30 sunscreen applied each morning. All products will be applied after facial cleansing, and sunscreen will be used 15 minutes prior to outdoor exposure. The treatment duration is 2 weeks, during which participants will record application times and any adverse effects in a diary. Assessments will be conducted at baseline, and at weeks 1, 2, and 4 post-laser, including standardized facial photography, modified Melasma Area and Severity Index (mMASI), mexameter readings, dermoscopy, Wood's lamp examination, and the Post-Acne Hyperpigmentation Index (PAHPI). Erythema scores and subjective assessments (VAS) will be recorded 15 minutes after the laser procedure.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-60 years.
* Patients diagnosed with post-acne hyperpigmentation and melasma based on clinical examination and Wood's lamp evaluation, with Fitzpatrick skin types IV and V.
* Patients visiting the Dermatology and Venereology Outpatient Clinic and scheduled to undergo QS Nd:YAG 1064 nm low-fluence laser treatment.

Patients who are currently receiving or have received a priming regimen for at least two weeks prior to the laser procedure, consisting of either 2% hydroquinone cream or a serum containing Niacinamide 10%, Hyaluronic Acid, and HEPES.

- Willing to participate in the study and provide written informed consent after receiving a complete explanation of the study procedures.

Exclusion Criteria:

* Pregnant, breastfeeding, or currently taking oral contraceptives at the time of evaluation.
* History of systemic retinoid use within the past three months.
* History of or ongoing treatment for hormonal/endocrine disorders or other severe systemic illnesses.
* Currently undergoing immunosuppressive therapy.
* Difficulty adhering to treatment protocols.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of Subjective Pain Evaluation | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  Assessed using Visual Analog Scale (VAS). Scale range is 0-10, 0 indicates no pain and 10 indicates severe pain
Change of Eryhtema Score | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  Based on Clinical Erythema Assessment Scale. Scale range is 0-4, 0 indicates no erythema and 4 indicates severe erythema
Change of Melasma Severity based on modified Melasma Severity Index (mMASI) score | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  the range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24). improvement occurs if the mMASI score decreases by <50% from the previous visit worsening if score persists or mMASI Score Increase >50%
Change of the Post-Acne Hyperpigmentation Index (PAHPI) score | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  On physical examination, the severity of post-inflammatory hyperpigmentation in patients with acne vulgaris was assessed using the Post-Acne Hyperpigmentation Index (PAHPI). The PAHPI score ranges from 6 to 22, with a score of 6 indicating mild post-acne hyperpigmentation and a score of 22 indicating severe post-acne hyperpigmentation.
Change of Melasma Severity based on Dermoscopy | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  based on Dermoscopy Telangiectasis score assessment using a 5-point dermoscopy-scale: 0 = No visible capillaries. 1 = Elongated capillaries accompanied by dilation, not visible to the naked eye. 2 = Moderate telangiectasis that is beginning to be visible to the naked eye. 3 = Severe telangiectasis characterized by reduced capillary loops. 4 = Very severe telangiectasis characterized by dilatation and loss of capillary loops.
Change of Melasma Severity based on Wood's Lamp | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  Epidermal Type/ Dermal Typed/ Mixed Typed
Change of Melanin Index Based on Mexameter | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  improves if there is a decrease in melanin levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in melanin levels or there is a decrease of <50%
Change of Erytema Index Based on Mexameter | baseline; 1 weeks post QS-Nd:YAG 1064 nm low-fluence laser; 2 weeks post QS-Nd:YAG 1064 nm low-fluence laser and 4 weeks post QS-Nd:YAG 1064 nm low-fluence laser
  improves if there is a decrease in Erytema levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in erythema levels or there is a decrease of <50%

CONTACTS AND LOCATIONS:
Locations (1):
- Gatot Soebroto Central Army Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided